CLINICAL TRIAL: NCT07406334
Title: A Phase 1, Observer-Blind, Randomized, Active Controlled Trial to Evaluate the Safety and Reactogenicity of an Investigational Pneumococcal Vaccine in Toddlers 12 To 15 Months of Age Receiving a Single Booster Dose
Brief Title: A Trial to Evaluate the Safety and Reactogenicity of an Investigational Pneumococcal Vaccine in Toddlers 12 to 15 Months of Age Receiving a Single Booster Dose
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 221546
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pneumonia, Bacterial
Keywords: Pneumococcal Vaccine; Phase 1; Pediatric; Booster dose
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is an observer-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pn-MAPS30plus Group (Experimental): Participants receive a single dose of Pn-MAPS30plus on Day 1.
  Interventions: Biological: Pn-MAPS30plus
- PCV20 Group (Active Comparator): Participants receive a single dose of PCV20 on Day 1.
  Interventions: Combination Product: PCV20

INTERVENTIONS:
Biological: Pn-MAPS30plus — Pn-MAPS30plus vaccine will be administered intramuscularly.
  Arms: Pn-MAPS30plus Group
Combination Product: PCV20 — PCV20 vaccine will be administered intramuscularly.
  Arms: PCV20 Group

SUMMARY:
The main purpose of this study is to assess the safety and reactogenicity of a single dose of the new pneumococcal vaccine (called Pn-MAPS30plus) in toddlers who have previously completed a two-dose primary vaccination series with PCV used in local immunization program. PCV20 will be used as a comparator for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants' parent(s)/Legally acceptable representative [LAR(s)] who, in the opinion of the investigator, can and will comply with all protocol requirements.
2. Written or witnessed/thumb printed informed consent obtained from the participants' parent(s)/LAR(s) prior any study-specific procedure is performed.
3. A male or female between, and including, 12 to15 Months of age at the time of the study intervention administration.
4. Healthy participants or medically stable patients as established by medical history and clinical examination before entering the study.
5. To the best knowledge of the participant's parent(s)/LAR(s), the child has been eligible for pneumococcal vaccination and has completed a 2-dose primary series with PCV10.

Exclusion Criteria:

1. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
2. Hypersensitivity to latex.
3. History of microbiologically proven Invasive pneumococcal Disease (IPD).
4. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
5. Major congenital defects, as assessed by the investigator.
6. Recurrent history or uncontrolled neurological disorders or any neuroinflammatory condition, congenital neurological conditions, encephalopathies, or seizures.
7. Condition that in the judgment of the investigator would make intramuscular injection unsafe.
8. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
9. Use of any investigational or non-registered product (drug, vaccine, or invasive medical device) during the period beginning 30 days before the dose of study intervention(s), or their planned use during the trial period.
10. Previous vaccination with any pneumococcal vaccine other than PCV10.
11. Previous receipt of more than 2 pneumococcal vaccine doses (primary series or booster).
12. Planned administration/administration of any inactivated or otherwise non-live vaccine in the period starting 14 days before and ending 14 days after the dose of study intervention administration or planned administration/administration of any live vaccine in the period starting 28 days before and ending 28 days after the dose of study intervention administration, with the exception of inactivated influenza vaccine which may be administered but must be given at least 7 days before or 15 days after receipt of any study intervention.
13. Receipt of blood or plasma products or immunoglobulins, from 90 days before study intervention administration, or planned receipt up to 30 days of study intervention administration.
14. Chronic administration of immune-modifying drugs and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

    * For corticosteroids: prednisone equivalent ≥0.5 mg/kg/day (maximum 20 mg/day) within 90 days prior for pediatric participants.
    * Inhaled and topical steroids are allowed.
15. Concurrent participation in another clinical study in which the participant has been or will be exposed to an investigational or non-investigational intervention.
16. Any child of trial personnel or their immediate dependents, family, or household members.
17. Child in care.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Administration site Adverse Events (AEs) | Day 1 to Day 7
  The AEs considered are tenderness, redness, and swelling at the administration site.
Number of Participants with Solicited Systemic Adverse Events (AEs) | Day 1 to Day 7
  The AEs considered are fever, irritability, loss of appetite and somnolence (sleepiness/drowsiness).
Number of Participants with Unsolicited AEs | Day 1 to Day 30
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Number of Participants with Serious AEs (SAEs), Adverse Events of Special Interest (AESIs) and AEs Leading to Withdrawal | Day 1 up to trial end (Month 6)
Number of Participants with Hematological and Biochemical Laboratory Abnormalities | On Day 8 compared to Day 1 (pre-vaccination)

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf